CLINICAL TRIAL: NCT00681161
Title: Autonomic Function in Obstructive Sleep Apnea (OSA)
Brief Title: Autonomic Function in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Amanda Peltier, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K23NS056009 (NIH); 1K23NS056009-01A1 (NIH)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; OSA; diabetes; pre-diabetic condition; obesity; blood glucose; continuous positive airway pressure; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus; Obesity | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other)
  Interventions: Other: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Other: continuous positive airway pressure (CPAP) — Standard of care treatment for OSA, requires a mask attached by tubing to a device providing continuous pressure of air at a given cm of water pressure, acting as a splint to open airway at night to relieve obstruction.

SUMMARY:
The purpose of this study is to determine if obstructive sleep apnea (OSA) causes autonomic dysfunction independent of its effects on hyperglycemia.

DETAILED DESCRIPTION:
The purpose of this study is to determine if obstructive sleep apnea (OSA)-a condition in which respiration and oxygenation are affected during sleep-can cause abnormal autonomic function and blood sugar (glucose) processing, which could lead to diabetes, or pre-diabetic conditions. The autonomic system controls heart rate, blood pressure, breathing, and other functions of the body. OSA and diabetes are commonly found in overweight individuals and both can cause increased risk of heart disease and strokes. OSA can be treated using nasal continuous positive airway pressure (CPAP) which overcomes the obstruction to airflow that occurs in OSA.

In this study, the scientists hope to determine if individuals with OSA have an increased prevalence of undiagnosed diabetes or pre-diabetic conditions, and if autonomic abnormalities observed previously in OSA are more severe or more common in people with OSA and diabetes or pre-diabetic conditions.

Participants will undergo a sleep study and glucose studies to determine if they have sleep apnea and impaired fasting glucose, impaired glucose tolerance, or undiagnosed diabetes (collectively called impaired glucose regulation).

Individuals with sleep apnea with and without glucose abnormalities will be age and BMI matched, and will undergo further autonomic and peripheral nerve testing. Individuals without diabetes will be followed for one year of CPAP treatment for their sleep apnea-with visits at 3 month intervals to evaluate glucose and autonomic function. Individuals without sleep apnea or diabetes will also undergo autonomic and peripheral nerve testing. Participants will also complete questionnaires to assess their sleepiness and symptoms of autonomic function.

Results from this study will help researchers determine if abnormalities of autonomic function seen in people with OSA are caused by OSA or by coexistent impaired glucose regulation present in people with OSA. In addition, results from the study will show if CPAP treatment improves autonomic dysfunction by correcting breathing abnormalities, or by secondary improvement of glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80.
* BMI between 25 and 35.
* Symptoms strongly indicative of sleep apnea (loud snoring, witnessed apneas or history of OSA based on laboratory PSG within 3 months of screening, not currently using CPAP, oral appliances or other treatments for OSA)

Exclusion Criteria:

* History of previous treatment for OSA.
* History of diabetes.
* History of other disorders known to affect autonomic function (e.g. Parkinson's disease, peripheral neuropathy of any cause, or requiring medications known to affect autonomic function that cannot be stopped safely for 48 hours).
* No evidence of peripheral neuropathy on examination, negative laboratory tests for common causes of neuropathy (B12, Thyroid stimulating hormone, serum protein electrophoresis).
* Inability to cooperate with testing, or to undergo testing (individuals with irregular heart rhythms, significant lung disease, previous LASIK procedure, unable to stop hypertensive medications for 48 hours).
* Medications affecting glucose levels, hypoglycemic agents, high dose thiazide diuretics, beta blocking agents.
* Pregnant or lactating females.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
blood glucose level, composite autonomic system score (CASS), homeostasis assessment model (HOMA), insulin sensitivity index (ISI) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amanda C. Peltier, MD, MS, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Peltier AC, Bagai K, Artibee K, Diedrich A, Garland E, Elasy T, Shi Y, Wang L, Feldman EL, Robertson D, Malow BA. Effect of mild hyperglycemia on autonomic function in obstructive sleep apnea. Clin Auton Res. 2012 Feb;22(1):1-8. doi: 10.1007/s10286-011-0131-9. Epub 2011 Jul 28. PMID 21796355